CLINICAL TRIAL: NCT05116046
Title: A PHASE 2 OPEN LABEL EXTENSION STUDY TO ASSESS THE LONG-TERM SAFETY, TOLERABILITY, PHARMACOKINETICS AND EFFICACY OF RECIFERCEPT IN CHILDREN WITH ACHONDROPLASIA
Brief Title: Continuation Study of Long-term Safety, Tolerability, Pharmacokinetics and Efficacy of Recifercept in Achondroplasia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated due to lack of efficacy at any of the tested doses on 18th November 2022. The decision to terminate the study is not related to a safety concern.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C4181008; 2021-003149-39 (EudraCT Number)
Record Dates: First submitted 2021-10-18; First posted 2021-11-10 (Actual); Results first posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Achondroplasia
Keywords: achondroplasia; dwarfism; bone diseases, development; bone diseases; Musculoskeletal Diseases; Osteochondrodysplasias; Genetic Diseases, Inborn; Skeletal Dysplasia
MeSH Terms: conditions — Achondroplasia; Dwarfism; Bone Diseases; Musculoskeletal Diseases; Osteochondrodysplasias; Genetic Diseases, Inborn; Mucopolysaccharidosis IV

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low Dose (Experimental): Low Dose
  Interventions: Biological: Recifercept
- Medium Dose (Experimental): Medium Dose
  Interventions: Biological: Recifercept
- High Dose (Experimental): High Dose
  Interventions: Biological: Recifercept

INTERVENTIONS:
Biological: Recifercept — Recifercept

SUMMARY:
All participants who completed the prior study to assess long-term safety, tolerability, pharmacokinetics and efficacy, and in the opinion of the investigator, continue to have a positive risk:benefit profile, will be offered to enroll in this open-label extension (OLE) study for up to an additional 24 months of treatment.

Approximately 63 participants will be offered to continue at the previously received dose of Recifercept either

Low Dose Medium Dose High Dose

or at the therapeutic dose once it is identified.

Participants will attend the clinic monthly for 24 months. Assessments include safety, blood sampling, physical examination, vital signs, anthropometric body measurements & patient/caregiver quality of life questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants between the ages of >15 months to <12 years inclusive, at Visit 1 (Screen 1).
* Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests lifestyle considerations and other study procedures.
* Completed the C4181005 Phase 2 study.
* Able to stand independently for height measurements (if ≥2 years of age at enrollment).

Exclusion Criteria:

* Presence of co-morbid conditions or circumstances that, in the opinion of the investigator, would affect interpretation of growth data or ability to complete the trial procedures.
* Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* Presence of severe obesity (body mass index (BMI) >95th percentile on Hoover-Fong BMI charts) [Hoover-Fong et al, 2008].
* Known closure of long bone growth plates (cessation of height growth).
* Body weight >45 kg.
* History of hypersensitivity to study intervention or any excipients.
* History of any prior treatment with human growth hormone or related products (including insulin-like growth factor 1 [IGF-1]).
* History of receipt of any treatment that are known to potentially affect growth (including oral steroids >5 days in the last 6 months, high dose inhaled corticosteroids (>800 mcg/day beclometasone equivalent) and medication for attention deficit hyperactivity disorder).
* History of limb lengthening surgery (defined as distraction osteogenesis/Ilizarov/callostasis technique following submetaphyseal osteotomy to extend bone length).
* Any limb lengthening/corrective orthopaedic surgery planned at any point during the trial period.
* Less than 6 months since fracture or surgical procedure of any bone determined from the screening visit date.
* Presence of any internal guided growth plates/devices.
* History of removal of internal guided growth plates/devices within less than 6 months.
* History of receipt of any other (except recifercept) investigational product for achondroplasia or that may affect growth/interpretation of growth parameters.
* History of receipt of an investigational drug (not for achondroplasia/growth affecting) within the last 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of study intervention used in this study (whichever is longer).

Ages: 15 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2021-12-24 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2023-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (13):
- United States (6):
  - Ocean Sleep Medicine, Irvine, California
  - Long Beach Memorial Medical Center, Long Beach, California
  - MemorialCare Sleep Disorders Center at Long Beach Memorial Medical Center, Long Beach, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Nemours Children's Hospital, Delaware, Wilmington, Delaware
  - Texas Childrens Hospital/Baylor College of Medicine, Houston, Texas
- Murdoch Children's Research Institute, Parkville, Victoria, Australia
- Belgium (2):
  - UZ Leuven - Center of Human Genetics, Leuven, Flanders
  - Antwerp University Hospital, Edegem
- Bispebjerg Hospital, Copenhagen, Denmark
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS Università Cattolica del Sacro Cuore, Roma, Italy
- Centro Hospitalar e Universitário de Coimbra - Hospital Pediátrico, Coimbra, Portugal
- Hospital Vithas San Jose, Vitoria-Gasteiz, Alava, Spain

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4181008

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants aged greater than or equal to (>=)15 months to 12 years (inclusive) diagnosed with achondroplasia from study C4181005 (NCT04638153) were enrolled in this extension study.
Pre-assignment Details: A total of 35 participants were enrolled and assigned to study treatment.
Groups:
- Recifercept 1 Milligram Per Kilogram (mg/kg) Once Weekly: Participants with achondroplasia who completed study C4181005 (NCT04638153) received recifercept 1 mg/kg once weekly via the subcutaneous route for up to 24 months.
- Recifercept 2 mg/kg Twice Weekly: Participants with achondroplasia who completed study C4181005 (NCT04638153) received recifercept 2 mg/kg twice weekly via the subcutaneous route for up to 24 months.
- Recifercept 1.5 mg/kg Once Daily: Participants with achondroplasia who completed study C4181005 (NCT04638153) received recifercept 1.5 mg/kg once daily via the subcutaneous route for up to 24 months.
Period: Overall Study
Arm/Group | Recifercept 1 Milligram Per Kilogram (mg/kg) Once Weekly | Recifercept 2 mg/kg Twice Weekly | Recifercept 1.5 mg/kg Once Daily
Started | 16 | 17 | 2
Completed | 0 | 0 | 0
Not Completed | 16 | 17 | 2
Not completed — Withdrawal by parent/guardian | 2 | 1 | 1
Not completed — Study terminated by sponsor | 14 | 16 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all participants who received at least 1 dose of recifercept. Participants were analyzed according to the dose they actually received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Recifercept 1 Milligram Per Kilogram (mg/kg) Once Weekly | Recifercept 2 mg/kg Twice Weekly | Recifercept 1.5 mg/kg Once Daily | Total
Number analyzed (Participants) | 16 | 17 | 2 | 35
Age, Continuous [Mean (Standard Deviation); unit: Years] | 7.5 (2.66) | 6.6 (2.50) | 9.5 (0.71) | 7.2 (2.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 2 | 20
  Male | 7 | 8 | 0 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 1 | 3
  Not Hispanic or Latino | 14 | 17 | 1 | 32
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 14 | 17 | 2 | 33
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs) and Severe AEs
Description: An AE was any untoward medical occurrence that did not necessarily have a causal relationship with study treatment. TEAE was an AE that occurred after initiation of study treatment that was not present at the time of treatment start or an AE that increased in severity after the initiation of medication, if the event was present at the time of treatment start emerges. SAE was an AE resulting in any of the following outcomes or considered medically significant: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly or birth defect. Severe AEs were AEs that were medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated disabling, limiting self-care activities of daily living.
Time Frame: From first dose of study drug up to 28 days after last dose of study drug (maximum up to 11 months)
Population: FAS consisted of all participants who received at least one dose of recifercept. Participants were analyzed according to the dose they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Recifercept 1 Milligram Per Kilogram (mg/kg) Once Weekly | Recifercept 2 mg/kg Twice Weekly | Recifercept 1.5 mg/kg Once Daily
Number analyzed (Participants) | 16 | 17 | 2
Participants
  AEs | 9 | 11 | 0
  SAEs | 0 | 0 | 0

2. Primary Outcome: Change From Baseline in Height at Month 24
Description: Height was measured using anthropometric measurements. Anthropometric data was collected by appropriately trained individuals at the trial site and in accordance with the anthropometric measurement manual.
Time Frame: Baseline, Month 24
Population: Data was not collected as study was terminated based on sponsor discretion due to lack of efficacy at any of the tested doses. The decision to terminate the study was not related to a safety concern.
Arm/Group | Recifercept 1 Milligram Per Kilogram (mg/kg) Once Weekly | Recifercept 2 mg/kg Twice Weekly | Recifercept 1.5 mg/kg Once Daily
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Clearance (CL/F) of Recifercept
Description: Clearance of a drug was a measure of the rate at which a drug is metabolised or eliminated by normal biological processes.
Time Frame: Predose on Day 91, 181, 271, 361 and 451.
Population: as for outcome 2
Arm/Group | Recifercept 1 Milligram Per Kilogram (mg/kg) Once Weekly | Recifercept 2 mg/kg Twice Weekly | Recifercept 1.5 mg/kg Once Daily
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Change From Baseline in Sitting Height to Standing Height Ratio at Months 3, 6, 9
Description: Sitting height to standing height ratio was calculated based upon the anthropometric measurements. Anthropometric data was collected by appropriately trained individuals at the trial site and in accordance with the anthropometric measurement manual.
Time Frame: Baseline and Months 3, 6, 9
Population: as for outcome 2
Arm/Group | Recifercept 1 Milligram Per Kilogram (mg/kg) Once Weekly | Recifercept 2 mg/kg Twice Weekly | Recifercept 1.5 mg/kg Once Daily
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Change From Baseline in Arm Span to Height/Length Difference at Months 3, 6, 9
Description: Height and length difference was calculated with anthropometric measurements. Anthropometric data was collected by appropriately trained individuals at the trial site and in accordance with the anthropometric measurement manual.
Time Frame: Baseline and Months 3, 6, 9
Population: as for outcome 2
Arm/Group | Recifercept 1 Milligram Per Kilogram (mg/kg) Once Weekly | Recifercept 2 mg/kg Twice Weekly | Recifercept 1.5 mg/kg Once Daily
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Change From Baseline in Knee Height to Lower Segment Ratio at Months 3, 6, 9
Description: Knee height was defined as the distance from the sole of the foot to the most anterior surface of the femoral condyles of the thigh (medial being more anterior), with the ankle and knee each flexed to a 90-degree angle. Lower segment of the leg included tibia and foot height
Time Frame: Baseline and Months 3, 6, 9
Population: as for outcome 2
Arm/Group | Recifercept 1 Milligram Per Kilogram (mg/kg) Once Weekly | Recifercept 2 mg/kg Twice Weekly | Recifercept 1.5 mg/kg Once Daily
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Change From Baseline in Occipito-Frontal Circumference at Months 3, 6, 9
Description: Occipito-frontal circumference was measured by anthropometric measurements. It was measured over the most prominent part on the back of the head (occiput) and just above the eyebrows (supraorbital ridges).
Time Frame: Baseline and Months 3, 6, 9
Population: as for outcome 2
Arm/Group | Recifercept 1 Milligram Per Kilogram (mg/kg) Once Weekly | Recifercept 2 mg/kg Twice Weekly | Recifercept 1.5 mg/kg Once Daily
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Change From Baseline in Occipito-Frontal Distance to Occipito-mid-Face Measurements Ratio at Months 3, 6, 9
Description: Occipito-frontal circumference was measured by anthropometric measurements. Anthropometric data was collected by appropriately trained individuals at the trial site and in accordance with the anthropometric measurement manual.
Time Frame: Baseline, Months 3, 6, 9
Population: as for outcome 2
Arm/Group | Recifercept 1 Milligram Per Kilogram (mg/kg) Once Weekly | Recifercept 2 mg/kg Twice Weekly | Recifercept 1.5 mg/kg Once Daily
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Change From Baseline in Z-Score for Occipito-frontal Circumference, Arm Span, Sitting Height and Skull Morphology at Months 3, 6, 9
Description: The Z-score described how many standard deviations a given measurement lies above or below a size or age-specific population mean. A Z-score above the population mean indicates a positive value, whereas a Z-score below the population mean indicates a negative value. The greater the deviation of the Z-score from zero (in a positive or negative direction), the greater the magnitude of deviation from the mean.
Time Frame: Baseline, Months 3, 6, 9
Population: as for outcome 2
Arm/Group | Recifercept 1 Milligram Per Kilogram (mg/kg) Once Weekly | Recifercept 2 mg/kg Twice Weekly | Recifercept 1.5 mg/kg Once Daily
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Change From Baseline in Fixed Flexion Angles at Elbow at Months 3, 6, 9
Description: Fixed Flexion Angles was measured by anthropometric measurements. Anthropometric data was collected by appropriately trained individuals at the trial site and in accordance with the anthropometric measurement manual.
Time Frame: Baseline, Months 3, 6, 9
Population: as for outcome 2
Arm/Group | Recifercept 1 Milligram Per Kilogram (mg/kg) Once Weekly | Recifercept 2 mg/kg Twice Weekly | Recifercept 1.5 mg/kg Once Daily
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Change From Baseline in Body Mass Index (BMI) at Months 3, 6, 9
Time Frame: Baseline, Months 3, 6, 9
Population: as for outcome 2
Arm/Group | Recifercept 1 Milligram Per Kilogram (mg/kg) Once Weekly | Recifercept 2 mg/kg Twice Weekly | Recifercept 1.5 mg/kg Once Daily
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Change From Baseline in Waist to Chest Circumference Ratio at Months 3, 6, 9
Time Frame: Baseline, Months 3, 6, 9
Population: as for outcome 2
Arm/Group | Recifercept 1 Milligram Per Kilogram (mg/kg) Once Weekly | Recifercept 2 mg/kg Twice Weekly | Recifercept 1.5 mg/kg Once Daily
Number analyzed (Participants) | 0 | 0 | 0

13. Secondary Outcome: Number of Participants With Clinically Meaningful Findings in Laboratory Test Parameters Through the Study
Description: Laboratory parameters that were assessed included lymphocytes, neutrophils, eosinophils, monocytes and potassium. Clinically significant abnormal laboratory findings were determined based on investigator's decision.
Time Frame: From baseline up to end of study/early termination (for a maximum duration of 11 months)
Population: FAS included all participants who were planned to receive at least one dose of recifercept. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.'
Measure: Count of Participants; unit: Participants
Arm/Group | Recifercept 1 Milligram Per Kilogram (mg/kg) Once Weekly | Recifercept 2 mg/kg Twice Weekly | Recifercept 1.5 mg/kg Once Daily
Number analyzed (Participants) | 15 | 16 | 2
Participants
  Hematology: Lymphocytes | 0 | 1 | 0
  Hematology: Neutrophils | 0 | 1 | 0
  Hematology: Eosinophils | 1 | 3 | 0
  Hematology: Monocytes | 2 | 0 | 0
  Chemistry: Potassium | 2 | 1 | 0

14. Secondary Outcome: Number of Participants With Clinically Significant Findings in Vital Signs Through the Study
Description: Absolute values and changes from baseline in supine systolic and diastolic blood pressure, oral temperature, and pulse rate were planned to be summarized by treatment in accordance with the sponsor reporting standards. Clinically significant abnormal laboratory findings were those which were not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
Time Frame: From baseline up to end of study/early termination (for a maximum duration of 11 months)
Population: FAS included all participants who were planned to receive at least one dose of recifercept.
Measure: Count of Participants; unit: Participants
Arm/Group | Recifercept 1 Milligram Per Kilogram (mg/kg) Once Weekly | Recifercept 2 mg/kg Twice Weekly | Recifercept 1.5 mg/kg Once Daily
Number analyzed (Participants) | 16 | 17 | 2
Participants | 0 | 0 | 0

15. Secondary Outcome: Number of Participants With Clinically Significant Findings in Physical Examination Through the Study
Description: A complete physical examination included cardiovascular, respiratory, gastrointestinal systems, and skin. Height and weight will also be measured and recorded as part of the anthropometric measurements collected. Anthropometric data was collected by appropriately trained individuals at the trial site and in accordance with the anthropometric measurement manual.
Time Frame: From baseline up to end of study/early termination (for a maximum duration of 11 months)
Population: FAS included all participants who were planned to receive at least one dose of recifercept.
Measure: Count of Participants; unit: Participants
Arm/Group | Recifercept 1 Milligram Per Kilogram (mg/kg) Once Weekly | Recifercept 2 mg/kg Twice Weekly | Recifercept 1.5 mg/kg Once Daily
Number analyzed (Participants) | 16 | 17 | 2
Participants | 0 | 0 | 0

16. Secondary Outcome: Number of Participants With Positive Anti-Drug Antibodies (ADA)
Time Frame: From Month 3 up to end of study/early termination (up to Month 11)
Population: FAS included all participants who were planned to receive at least one dose of recifercept.
Measure: Count of Participants; unit: Participants
Arm/Group | Recifercept 1 Milligram Per Kilogram (mg/kg) Once Weekly | Recifercept 2 mg/kg Twice Weekly | Recifercept 1.5 mg/kg Once Daily
Number analyzed (Participants) | 16 | 17 | 2
Participants | 12 | 15 | 2

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 28 days after last dose of study drug (maximum up to 11 months)
Groups:
- Recifercept 1 mg/kg Once Weekly: Participants with achondroplasia who completed study C4181005 (NCT04638153) received recifercept 1 mg/kg once weekly via the subcutaneous route for up to 24 months.
Arm/Group | Recifercept 1 mg/kg Once Weekly | Recifercept 2 mg/kg Twice Weekly | Recifercept 1.5 mg/kg Once Daily
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/17 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/17 | 0/2
Other Adverse Events (participants affected / at risk) | 9/16 | 11/17 | 0/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Recifercept 1 mg/kg Once Weekly (N=16) | Recifercept 2 mg/kg Twice Weekly (N=17) | Recifercept 1.5 mg/kg Once Daily (N=2)
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0
Eustachian tube dysfunction (Ear and labyrinth disorders) | 0 | 1 | 0
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 | 1 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 0
Injection site rash (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0
COVID-19 (Infections and infestations) | 2 | 0 | 0
Conjunctivitis (Infections and infestations) | 1 | 0 | 0
Injection site haematoma (General disorders) | 1 | 0 | 0
Ear infection (Infections and infestations) | 1 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 2 | 1 | 0
Nasopharyngiti (Infections and infestations) | 3 | 1 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 0
Otitis externa (Infections and infestations) | 0 | 1 | 0
Otitis media (Infections and infestations) | 1 | 1 | 0
Otitis media acute (Infections and infestations) | 1 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 4 | 0
Skin candida (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Vaccination complication (Injury, poisoning and procedural complications) | 1 | 1 | 0
Blood phosphorous increased (Investigations) | 1 | 0 | 0
Blood urea increase (Investigations) | 1 | 0 | 0
Platelet count increased (Investigations) | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Nystagmus (Nervous system disorders) | 1 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 1 | 0
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 2 | 0

LIMITATIONS AND CAVEATS:
Data was not collected for efficacy endpoints as study was terminated early based on sponsor discretion due to lack of efficacy at any of the tested doses. The decision to terminate the study was not related to a safety concern.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-05-17): https://cdn.clinicaltrials.gov/large-docs/46/NCT05116046/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-28): https://cdn.clinicaltrials.gov/large-docs/46/NCT05116046/SAP_001.pdf